CLINICAL TRIAL: NCT02248038
Title: A Multicenter Randomized Clinical Trial on Laparoscopic Colorectal Cancer Surgery Compared With Open Surgery in China
Brief Title: A Multicenter Clinical Trial on Laparoscopic Colorectal Cancer Surgery Compared With Open Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cai Kailin (Other)
Collaborators: Huazhong University of Science and Technology (Other); Nanfang Hospital, Southern Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Cai Kailin, Associate chief physician of gastrointestinal surgery, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR-TRC-14004767; ChiCTR-TRC-14004767 (Registry Identifier: ChiCTR-TRC-14004767)
Record Dates: First submitted 2014-09-09; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open surgery (Active Comparator): Conventional procedure
  Interventions: Procedure: open surgery
- laparoscopic surgery (Experimental): Minimum invasive procedure
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: open surgery — Patients in this arm undergo radical resection of colon cancer in open surgery.Open surgery is a conventional technique for colorectal cancer patients.
  Other Names: open
  Arms: open surgery
Procedure: laparoscopic surgery — Patients in this arm undergo radical resection of colon cancer in laparoscopic surgery.Laparoscopic surgery is a new and minimum invasive technique for colorectal cancer patients.
  Other Names: laparoscopic
  Arms: laparoscopic surgery

SUMMARY:
The purpose of this study is to verify the 5-year disease free survival (DFS) of resectable colorectal cancer after laparoscopic surgery according to a Chinese Operative Standard was not inferior to open surgery.

DETAILED DESCRIPTION:
Study type：Interventional Study phase：Phase III Objectives of Study：to verify the 5-year DFS of resectable colorectal cancer after laparoscopic surgery according to a Chinese Operative Standard was not inferior to open surgery.

Study design：Randomized parallel control

ELIGIBILITY:
Inclusion Criteria:

1. informed consent
2. single colorectal adenocarcinoma, located at any segment of the colorectum with lower margin 5cm or more to the dental line
3. cTNM：colon cancer T1-4N1-2M0，rectal cancer T1-3N1-2M0，longest diameter no more than 6cm
4. age less than 80 years old
5. normal blood routine test and hepatic or renal function test
6. no gastrointestinal surgery history or chemotherapy, radiation, No complete obstruction.

Exclusion Criteria:

1. severe comorbidity such as heart attack or stroke, malignance in 5 years
2. can not tolerate to general anesthesia, pneumoperitoneum or surgery
3. pregnant or during breast-feeding period
4. attending other clinical trial involving therapy
5. cannot or disagree to attending the clinical trial

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
5 years diseases free survival rate | five years
5 years overall survival rate | five years

CONTACTS AND LOCATIONS:
Overall Officials: Guobin Wang, MD,PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Kaixiong Tao, MD,PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Kailin Cai, MD,PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Shi Wang, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China